CLINICAL TRIAL: NCT02792374
Title: Psychological Profile of Dental Patients. A Case Control Study
Brief Title: Psychological Profile of Dental Patients
Status: Completed | Type: Observational
Sponsor: Talebian, Alireza, M.D. (Individual)
Responsible Party: Principal Investigator, Talebian, Alireza, M.D., Dr, Talebian, Alireza, M.D.
Other Study IDs: 1818193574
Record Dates: First submitted 2016-05-26; First posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Indication for Modification of Patient Psychological Status
Keywords: Dental patients; Psychological Profile

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dental patients group: Psychological measurement is done when they refer to a dental clinic.
  Interventions: Other: Psychological Measurement
- Control group: Psychological measurement is done when they refer to a dental clinic.
  Interventions: Other: Psychological Measurement

INTERVENTIONS:
Other: Psychological Measurement — Measurement of psychological status in three levels: discrete symptom level, dimensional level, global level as measured by the scale
  Other Names: psychological assessment of the subjects

SUMMARY:
The objective of this descriptive investigation was to evaluate the psychological profile of dental patients in three levels: global level, the dimensional level, and the discrete symptom level and to compare it with a control group.

DETAILED DESCRIPTION:
Many people is afraid of dental treatment specially local anesthesia and do not refer to dental clinics until they are obliged due to dental pain. There are so many articles in the literature about dental phobia and fear of anesthetic injection. Due to these evidences, dental people are supposed to show elevated psychological dimensions such as anxiety, and somatization.

We are going to know which psychological dimensions of dental patients may be elevated when they refer to dental clinics.

ELIGIBILITY:
Inclusion Criteria:

Must:

be ≥ 18 years old and have high school degree or higher

Exclusion Criteria:

insufficient verbal capacity to comprehend the items of the questionnaire.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who referred to a dental office in Isfahan city, Iran. The chief complaints of them were not the same.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2012-01; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Nine psychological dimensions measured using a self-administered scale (SCL-90-R) | through study completion, an average of 1 year
  The subjects are supposed to consider the last week and answer all questions of psychological questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Talebian, PhD, Principal Investigator — Cheif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eli I, Baht R, Kozlovsky A, Rosenberg M. The complaint of oral malodor: possible psychopathological aspects. Psychosom Med. 1996 Mar-Apr;58(2):156-9. doi: 10.1097/00006842-199603000-00010. PMID 8849633
- See also: Click here for more information about this study: The complaint of oral malodor — http://journals.lww.com/psychosomaticmedicine/Abstract/1996/03000/The_Complaint_of_Oral_Malodor__Possible.10.aspx